CLINICAL TRIAL: NCT03007420
Title: A Prospective Controlled Treatment Trial for Post-Traumatic Headaches
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated prematurely by the study Principal Investigator due to slow patient recruitment.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Pradeep Dinakar, MD, MS, FAAP, Assistant Professor of Anesthesiology, Harvard Medical School; Staff Physician, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00025021
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Post-Traumatic Headaches
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Occipital Nerve Block (Experimental): After enrollment in the study, patients will be randomized (but not blinded) to receive either an occipital nerve block or a cervical medial branch block. These are injections of anti-inflammatory medications (steroids) and numbing medications (local anesthetics -lidocaine) in nerves located at the back of the head and neck. If patients exhibit a > or = 50% pain reduction on receiving the block evaluated after four weeks, then they may continue to receive blocks as needed, but not more than one every three months.
  If patients exhibit < 50% pain reduction, the patient will be treated as per the clinician's judgment with the possibility of a cross over to the other treatment option.
  Interventions: Drug: Occipital Nerve Block (ONB) using lidocaine and dexamethosone
- Cervical Medial Branch Block (Experimental): After enrollment in the study, patients will be randomized (but not blinded) to receive either an occipital nerve block or a cervical medial branch block. These are injections of anti-inflammatory medications (steroids) and numbing medications (local anesthetics -lidocaine) in nerves located at the back of the head and neck. If patients exhibit a > or = 50% pain reduction on receiving the block evaluated after four weeks, then they may continue to receive blocks as needed, but not more than one every three months.
  If patients exhibit < 50% pain reduction the patient will be treated as per the clinician's judgment with the possibility of a cross over to the other treatment option.
  Interventions: Drug: Cervical Medial Branch Block (CMBB) using lidocaine and dexamethosone

INTERVENTIONS:
Drug: Occipital Nerve Block (ONB) using lidocaine and dexamethosone — Patients enrolled in the study will be randomized to receive either an ONB or a CMBB. The assignment of the procedure will be randomized however neither the patients nor the investigator will be blinded to the procedure. Patients randomized to receive an ONB will receive the block with dexamethasone 2mg (steroid) each site with 3ml 1% lidocaine (local anesthetic), for a total of two sites.
  Arms: Occipital Nerve Block
Drug: Cervical Medial Branch Block (CMBB) using lidocaine and dexamethosone — Patients enrolled in the study will be randomized to receive either an ONB or a CMBB. The assignment of the procedure will be randomized however neither the patients nor the investigator will be blinded to the procedure. Patients randomized to receive CMBB will receive the block with dexamethasone 1.5mg (steroid) each site with 2 ml 1% lidocaine (local anesthetic), for a total of three sites on each side.
  Arms: Cervical Medial Branch Block

SUMMARY:
Post-traumatic headaches (PTH) are the most common complaint after traumatic brain injury, possibly generated by a number of stressors to the trigeminovascular and cervical plexus networks, including inflammation of the high cervical facet joints, traumatic cranial neuralgias, migraines, and myofascial injuries. To date, no treatment guidelines exist for PTH management except for conservative modalities, such as cognitive rest, physical therapy, and neuropathic pain medications, all of which have minimal evidence to support them.

The investigators propose a randomized, controlled, clinical trial and prospective follow-up study to evaluate the effect of invasive procedures such as occipital nerve block (ONB) and cervical medial branch block (CMBB) in the management of PTH.

Adolescents and adults (14-45 years of age) will be recruited from Boston Children's Hospital and Beth Israel Deaconess Medical Center Pain clinics, Concussion clinics and Headache clinics.

DETAILED DESCRIPTION:
Headaches and neck pain following a concussion are potentially treatable and resolve over time. Nerve blockade may enhance the recovery of appropriate neural circuits involved in the pathophysiology of a chronic headache. Currently, no evidence-based guidelines exist for treatment of PTH. Adoption of "brain rest" for 1-2 weeks, followed by gradual return to activity and avoiding "second-impact syndrome" are current practice. The use of medications controlling neuropathic pain is of partial benefit for some. Adverse effects like sedation, mood changes, cardiac side effects of pharmacologic agents are often not compatible with the demands of athletics. For those patients where sports performance is paramount, they may therefore not be able to tolerate regular medications. The incidence of chronic post-concussive headaches (> 3 months) at one year is 8.4% - 35% and at four years is up to 25%. Therefore, patients can have a significant disability from their post-traumatic headaches for many years after their injury. Without appropriate treatment, these headaches can remain as chronic headaches. Over-the-counter and other symptomatic medication overuse can exacerbate and prolong PTH significantly, secondary to rebound headaches. Successful treatment is essential since PTH limits return to sports as well as more general activities of living, such as work and school. Most interventions currently in use partially help and take several weeks to months for a noticeable benefit. PTH interventions, including ONB and CMBB, are employed in the treatment of primary headache disorders and neck pain from cervical arthritis and may provide more improved, faster and more sustained pain relief in many patients. Also, given that most of the action of the nerve blocks is local, there are significantly fewer side effects than in more standard headache medications. Injections that use corticosteroids may be beneficial in a post-traumatic headache by reducing inflammation and therefore mechanical allodynia. Injection of corticosteroids in the cervical facet joint area has shown up to 13 months of pain relief. This prolonged effect may be secondary to central pain modulation. Ultimately, nerve blocks may be a more effective and efficient post-traumatic headache given the onset of effect and the minimal side effects.

To date, there have been no prospective studies of procedural treatments for medically refractory PTH and none in the adolescent and young adult population in whom football injuries are common. Despite the frequent clinical practice of using ONB and CMBB for occipital neuralgia, cervical arthritis, and cervicogenic headaches, there has been no adequate scientific investigation into the use of these interventions for PTH. Given that PTH is typically felt to be secondary to an inflammatory reaction to trauma, the use of injection of corticosteroids may be more effective in PTH than in common headache disorders.

The investigators propose a randomized, prospective, controlled treatment trial to evaluate the efficacy of minimally invasive nerve block interventions (ONB and CMBB) as treatments for PTH and neck pain in adolescents and adults aged 14-45 years of age with PTH.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 - 45 years
* History of post-traumatic headache or neck pain following a concussion or head injury within the last 12 months
* Self-reported lack of meaningful benefit with at least one previous treatment trial. Previous treatment could include a migraine prophylactic medication, a neuropathic pain medication, a physical intervention, or a cognitive-behavioral intervention.

Exclusion Criteria:

* Significant underlying psychological concerns, as determined by study psychologist up on review of standardized assessment
* Lack of parental consent and child assent (if patient age <18 years) or lack of consent (if patient age >18 years). Unable to complete the questionnaire, based on parental or patient estimation of cognitive or language limitations

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share any IPD collected during the study with other researchers not included in the protocol.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were recruited from Boston Children's Hospital and Beth Israel Deaconess Medical Center. Eligibility Criteria included:
  * Age 14 - 45 years.
  * History of post-traumatic headache or neck pain following a concussion or head injury within the last 2 years.
  * Self-reported lack of meaningful benefit with at least one previous treatment trial.
Groups:
- Occipital Nerve Block; Cervical Medial Branch Block: After enrollment in the study, patients were randomized (but not blinded) to receive either an occipital nerve block or a cervical medial branch block. If patients exhibited a > or = 50% pain reduction on receiving the block evaluated after four weeks, they had an option to continue receiving blocks as needed, but not more than one every three months.
  If patients exhibited < 50% pain reduction, they were treated as per the clinician's judgment with the possibility of a cross over to the other treatment option.
Period: Overall Study
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Started | 8 | 8
Crossover | 3 | 2
Completed | 8 | 5
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: This study was terminated early due to slow patient recruitment. Given this, data has been analyzed for all patients enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (6) | 21 (7) | 22 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 1 | 4
Pain Score at Baseline [Median (Inter-Quartile Range); unit: units on a scale] — Pain Scores were assessed using the Numerical Rating Scale 0-10 with 0 being 'no pain' and 10 being 'worst pain imaginable'.
  units on a scale | 3.8 [2.5 to 5.6] | 4.9 [3.5 to 5.8] | 4.6 [2.7 to 5.8]
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Pain intensity was rated using the Numerical Rating Scale (NRS) of 0 to 10, with 0 indicating 'no pain' and 10 indicating the 'worst pain imaginable'.
Time Frame: One week, 1 month, 2 months, 3 months, 6months, 9 months, 12 months post-procedure
Population: 16 patients provided baseline pain score data that has been presented in the Baseline Demographics section. Post-procedure pain scores have been reported below.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 8 | 7
units on a scale
  Numerical Rating Scale at 1 week post procedure timepoint | 2.9 [1.5 to 4.7] | 3.7 [1.5 to 4.5]
  Numerical Rating Scale at 1 month post procedure time point: number analyzed (Participants) | 5 | 6
  Numerical Rating Scale at 1 month post procedure time point | 1 [0.4 to 2.4] | 1.6 [1 to 3.3]
  Numerical Rating Scale at 2 months post procedure time point: number analyzed (Participants) | 4 | 5
  Numerical Rating Scale at 2 months post procedure time point | 2.3 [1.3 to 4.6] | 5.2 [2 to 5.5]
  Numerical Rating Scale at 3 months post procedure time: number analyzed (Participants) | 6 | 4
  Numerical Rating Scale at 3 months post procedure time | 2.1 [1.2 to 3] | 1.7 [0 to 3.5]
  Numerical Rating Scale at 6 months post procedure time: number analyzed (Participants) | 5 | 3
  Numerical Rating Scale at 6 months post procedure time | 1.8 [1 to 4] | 0.8 [0.4 to 2.9]
  Numerical Rating Scale at 9 months post procedure time: number analyzed (Participants) | 5 | 2
  Numerical Rating Scale at 9 months post procedure time | 0 [0 to 3.5] | 3.6 [2.6 to 4.5]
  Numerical Rating Scale at 12 months post procedure time: number analyzed (Participants) | 3 | 2
  Numerical Rating Scale at 12 months post procedure time | 0.5 [0.3 to 0.6] | 3.4 [3 to 3.9]

2. Secondary Outcome: Migraine Disability Assessed Using the Migraine Disability Assessment (MIDAS)
Description: The Migraine Disability Assessment (MIDAS) is a self-administered standardized questionnaire to quantify headache-related disability.
  The MIDAS score ranges from 0 to 270. The higher the score on the MIDAS questionnaire, the greater the disability caused by headaches.
Time Frame: Baseline, 3 months, 6 months, 9 months, 12 months
Population: The Migraine Disability Assessment (MIDAS) is validated for patients 18 years and older only.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Occipital Nerve Block: After enrollment in the study, patients will be randomized (but not blinded) to receive either an occipital nerve block or a cervical medial branch block. These are injections of anti-inflammatory medications (steroids) and numbing medications (local anesthetics -lidocaine) in nerves located at the back of the head and neck. If patients exhibit a > or = 50% pain reduction on receiving the block evaluated after four weeks, then they may continue to receive blocks as needed, but not more than one every three months.
  If patients exhibit < 50% pain reduction, the patient will be treated as per the clinician's judgment with the possibility of a cross over to the other treatment option.
  Occipital Nerve Block (ONB) using lidocaine and dexamethosone: Patients enrolled in the study will be randomized to receive either an ONB or a CMBB. The assignment of the procedure will be randomized however neither the patients nor the investigator will be blinded to the procedure. Patients randomized to receive an ONB will receive the block with dexamethasone 2mg (steroid) each site with 3ml 1% lidocaine (local anesthetic), for a total of two sites.
- Cervical Medial Branch Block: After enrollment in the study, patients will be randomized (but not blinded) to receive either an occipital nerve block or a cervical medial branch block. These are injections of anti-inflammatory medications (steroids) and numbing medications (local anesthetics -lidocaine) in nerves located at the back of the head and neck. If patients exhibit a > or = 50% pain reduction on receiving the block evaluated after four weeks, then they may continue to receive blocks as needed, but not more than one every three months.
  If patients exhibit < 50% pain reduction the patient will be treated as per the clinician's judgment with the possibility of a cross over to the other treatment option.
  Cervical Medial Branch Block (CMBB) using lidocaine and dexamethosone: Patients enrolled in the study will be randomized to receive either an ONB or a CMBB. The assignment of the procedure will be randomized however neither the patients nor the investigator will be blinded to the procedure. Patients randomized to receive CMBB will receive the block with dexamethasone 1.5mg (steroid) each site with 2 ml 1% lidocaine (local anesthetic), for a total of three sites on each side.
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 5 | 5
units on a scale
  MIDAS Score at Baseline | 85 [53 to 94] | 159 [55 to 168]
  MIDAS Score at 3 months: number analyzed (Participants) | 3 | 3
  MIDAS Score at 3 months | 16 [12 to 59.5] | 43 [26 to 49.5]
  MIDAS Score at 6 months: number analyzed (Participants) | 2 | 3
  MIDAS Score at 6 months | 96 [68 to 124] | 5 [2.5 to 18.5]
  MIDAS Score at 9 months: number analyzed (Participants) | 2 | 1
  MIDAS Score at 9 months | 26.5 [26.5 to 26.75] | 60 [60 to 60]
  MIDAS Score at 12 months: number analyzed (Participants) | 2 | 1
  MIDAS Score at 12 months | 9 [4.5 to 13.5] | 39 [39 to 39]

3. Secondary Outcome: Pediatric Migraine Disability Assessment (PedMIDAS)
Description: The Pediatric Migraine Disability Assessment (PedsMIDAS) is a self-administered standardized questionnaire to quantify headache related disability.
  The PedsMIDAS score ranges from 0 to 240. The higher the score on the PedsMIDAS questionnaire, the greater the disability caused by headaches.
Time Frame: Baseline, 3 months, 6 months, 9 months, 12 months
Population: PedsMIDAS is only validated for patients for patients under the age of 18 years.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 3 | 3
units on a scale
  PedsMIDAS at Baseline | 227 [205 to 248] | 70 [42 to 151.5]
  PedsMIDAS at 3 months: number analyzed (Participants) | 3 | 1
  PedsMIDAS at 3 months | 23 [11.5 to 88.5] | 217 [217 to 217]
  PedsMIDAS at 6 months: number analyzed (Participants) | 3 | 0
  PedsMIDAS at 6 months | 16 [8 to 75] |
  PedsMIDAS at 9 months: number analyzed (Participants) | 3 | 1
  PedsMIDAS at 9 months | 9 [4.5 to 72] | 67 [67 to 67]
  PedsMIDAS at 12 months: number analyzed (Participants) | 1 | 1
  PedsMIDAS at 12 months | 0 [0 to 0] | 68 [68 to 68]

4. Secondary Outcome: Headache Severity Assessed by Migraine Disability Assessment (MIDAS)
Description: Self-administered questionnaire to quantify headache-severity using the following question:
  On a scale of 0 - 10, on average how painful were these headaches? (where 0=no pain at all, and 10=pain as bad as it can be)
Time Frame: Baseline, 3 months, 6 months, 9 months, 12 months
Population: The Migraine Disability Assessment (MIDAS) is validated for patients 18 years and older only.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 5 | 5
units on a scale
  MIDAS severity at baseline | 6 [5 to 7] | 6 [4 to 7]
  MIDAS severity at 3 months: number analyzed (Participants) | 3 | 3
  MIDAS severity at 3 months | 3 [3 to 4] | 3 [2.5 to 4]
  MIDAS severity at 6 months: number analyzed (Participants) | 2 | 3
  MIDAS severity at 6 months | 4.5 [3.25 to 5.75] | 4 [3 to 4.5]
  MIDAS severity at 9 months: number analyzed (Participants) | 2 | 1
  MIDAS severity at 9 months | 4 [3 to 5] | 6 [6 to 6]
  MIDAS severity at 12 months: number analyzed (Participants) | 2 | 1
  MIDAS severity at 12 months | 1 [0.5 to 1.5] | 4 [4 to 4]

5. Secondary Outcome: Headache Severity Assessed by the Pediatric Migraine Disability Assessment (PedMIDAS)
Description: Self-administered questionnaire to quantify headache-related disability
Time Frame: Baseline, 3 months, 6 months, 9 months, 12 months
Population: Although the investigators initially intended to assess headache severity using the PedsMIDAS questionnaire, it was discovered the specific headache severity assessment question was not included in the validated PedsMIDAS questionnaire. Consequently, we are unable to report data for this measure. Other alternate measures are reported. This was identified and reported as a minor deviation.
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Functional Disability Inventory Scores (FDI)
Description: The Functional Disability Inventory (FDI) was used to assess functional disability.
  The FDI is scored by summing the ratings for each of its 15 items, with scores ranging from 0 to 60.
  Higher scores indicate greater perceived functional disability.
Time Frame: Baseline, 3 months, 6 months, 9 months, 12 months
Population: The FDI is validated in patients under the age 18 years.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 3 | 3
units on a scale
  FDI Score at Baseline | 9 [9 to 18.5] | 18 [11 to 26.5]
  FDI Score at 3 months: number analyzed (Participants) | 3 | 1
  FDI Score at 3 months | 11 [5.5 to 19.5] | 30 [30 to 30]
  FDI Score at 6 months: number analyzed (Participants) | 3 | 0
  FDI Score at 6 months | 17 [8.5 to 22] |
  FDI Score at 9 months: number analyzed (Participants) | 3 | 1
  FDI Score at 9 months | 10 [5 to 16] | 14 [14 to 14]
  FDI Score at 12 months: number analyzed (Participants) | 1 | 1
  FDI Score at 12 months | 0 [0 to 0] | 4 [4 to 4]

7. Secondary Outcome: Pain Disability Index (PDI)
Description: The Pain Disability Index (PDI) was used to assess functional disability in adults.
  The PDI is scored by summing the ratings of seven different life domains, each scored on a scale of 0 to 10, with higher scores indicating greater pain-related disability.
  The total score can range from 0 to 70. A higher score reflects a greater impact of pain on daily activities.
Time Frame: Baseline, 3 months, 6 months, 9 months, 12 months
Population: The PDI is validated in patients 18 years of age or older.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 5 | 5
units on a scale
  PDI Score at Baseline | 30 [29 to 33] | 36 [11 to 37]
  PDI Score at 3 months: number analyzed (Participants) | 3 | 3
  PDI Score at 3 months | 19 [13.5 to 22] | 0 [0 to 7.5]
  PDI Score at 6 months: number analyzed (Participants) | 2 | 3
  PDI Score at 6 months | 16 [10.5 to 21.5] | 0 [0 to 11]
  PDI Score at 9 months: number analyzed (Participants) | 2 | 1
  PDI Score at 9 months | 2.5 [1.25 to 3.75] | 13 [13 to 13]
  PDI Score at 12 months: number analyzed (Participants) | 2 | 1
  PDI Score at 12 months | 6 [5.5 to 6.5] | 10 [10 to 10]

8. Secondary Outcome: World Health Organization Quality of Life - Brief Assessment (WHOQOL-BREF)
Description: The WHOQOL-BREF produces four domain scores (Physical health, Psychological, Social Relationships, and Environment) and two overall items (overall quality of life and general health). The scores range from 4-20 with higher scores indicating a better quality of life.
Time Frame: Baseline, 2 months, 3 months, 6 months, 9 months, 12 months
Population: WHOQOL-BREF is validated in adults 18 years of age or older.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 5 | 5
units on a scale
  WHOQOL-BREF Physical Health Scores at Baseline | 10.9 [9.7 to 11.4] | 12 [10.9 to 13.7]
  HOQOL-BREF Psychological Health Scores at Baseline | 11.3 [10.7 to 12] | 14 [12 to 15.3]
  HOQOL-BREF Social Relationship Scores at Baseline | 14.7 [12 to 16] | 14.7 [14.7 to 16]
  HOQOL-BREF Environment Scores at Baseline: number analyzed (Participants) | 5 | 4
  HOQOL-BREF Environment Scores at Baseline | 15.5 [15.5 to 16.5] | 15.3 [15 to 16]
  HOQOL-BREF Physical Health Scores at 2 months: number analyzed (Participants) | 3 | 4
  HOQOL-BREF Physical Health Scores at 2 months | 12.6 [12.6 to 12.9] | 12.6 [11.7 to 13.9]
  HOQOL-BREF Psychological Health Scores at 2 months: number analyzed (Participants) | 3 | 4
  HOQOL-BREF Psychological Health Scores at 2 months | 12 [10.7 to 12.7] | 13.3 [11.7 to 14.7]
  HOQOL-BREF Social Relationships Scores at 2 months: number analyzed (Participants) | 3 | 4
  HOQOL-BREF Social Relationships Scores at 2 months | 16 [15.3 to 16] | 13.3 [13 to 15]
  HOQOL-BREF Environment Scores at 2 months: number analyzed (Participants) | 3 | 4
  HOQOL-BREF Environment Scores at 2 months | 15.5 [15 to 15.8] | 16 [14.9 to 17.4]
  HOQOL-BREF Physical Health Scores at 3 months: number analyzed (Participants) | 3 | 2
  HOQOL-BREF Physical Health Scores at 3 months | 13.1 [12.9 to 13.1] | 13.7 [12.9 to 14.6]
  HOQOL-BREF Psychological Health Scores at 3 months: number analyzed (Participants) | 3 | 2
  HOQOL-BREF Psychological Health Scores at 3 months | 12.7 [12.7 to 12.7] | 15 [13.8 to 16.2]
  WHOQOL-BREF Social Relationship Scores at 3 months: number analyzed (Participants) | 3 | 2
  WHOQOL-BREF Social Relationship Scores at 3 months | 16 [14.7 to 16.7] | 16 [14 to 18]
  WHOQOL-BREF Environment Scores at 3 months: number analyzed (Participants) | 3 | 2
  WHOQOL-BREF Environment Scores at 3 months | 15.5 [15 to 16.8] | 18 [17 to 19]
  WHOQOL-BREF Physical Health Scores at 6 months: number analyzed (Participants) | 2 | 3
  WHOQOL-BREF Physical Health Scores at 6 months | 12 [11.4 to 12.6] | 13.1 [12.9 to 14]
  WHOQOL-BREF Psychological Health Scores at 6 months: number analyzed (Participants) | 2 | 3
  WHOQOL-BREF Psychological Health Scores at 6 months | 13 [12.8 to 13.7] | 14.7 [13.3 to 16]
  WHOQOL-BREF Social Relationship Scores at 6 months: number analyzed (Participants) | 1 | 3
  WHOQOL-BREF Social Relationship Scores at 6 months | 14.7 [14.7 to 14.7] | 16.5 [16.3 to 17.8]
  WHOQOL-BREF Environment Scores at 6 months: number analyzed (Participants) | 2 | 3
  WHOQOL-BREF Environment Scores at 6 months | 15.5 [15.3 to 15.8] | 16.5 [16.3 to 17.8]
  WHOQOL-BREF Physical Health Scores at 9 months: number analyzed (Participants) | 2 | 1
  WHOQOL-BREF Physical Health Scores at 9 months | 12.9 [12.1 to 13.6] | 12.6 [12.6 to 12.6]
  WHOQOL-BREF Psychological Health Scores at 9 months: number analyzed (Participants) | 2 | 1
  WHOQOL-BREF Psychological Health Scores at 9 months | 15 [14.8 to 15.2] | 12 [12 to 12]
  WHOQOL-BREF Social Relationship Scores at 9 months: number analyzed (Participants) | 0 | 1
  WHOQOL-BREF Social Relationship Scores at 9 months |  | 16 [16 to 16]
  WHOQOL-BREF Environment Scores at 9 months: number analyzed (Participants) | 2 | 1
  WHOQOL-BREF Environment Scores at 9 months | 16.3 [15.9 to 16.6] | 16 [16 to 16]
  WHOQOL-BREF Physical Health Scores at 12 months: number analyzed (Participants) | 2 | 1
  WHOQOL-BREF Physical Health Scores at 12 months | 14.6 [14.4 to 14.7] | 12 [12 to 12]
  WHOQOL-BREF Psychological Health Scores at 12 months: number analyzed (Participants) | 2 | 1
  WHOQOL-BREF Psychological Health Scores at 12 months | 15.3 [14.7 to 16] | 11.3 [11.3 to 11.3]
  WHOQOL-BREF Social Relationship Scores at 12 months: number analyzed (Participants) | 2 | 1
  WHOQOL-BREF Social Relationship Scores at 12 months | 14.7 [14 to 15.3] | 14.7 [14.7 to 14.7]
  WHOQOL-BREF Environment Scores at 12 months: number analyzed (Participants) | 2 | 1
  WHOQOL-BREF Environment Scores at 12 months | 16 [15.8 to 16.3] | 16 [16 to 16]

9. Secondary Outcome: Pediatric Quality of Life Assessment (PedsQL)
Description: The Pediatric Quality of Life Assessment (PedsQL) is a standardized questionnaire that assesses a pediatric patient's perceptions of health-related quality of life (HRQOL) with chronic health conditions using 4 domains (Physical, Emotional, Social, School Functioning).
  PedsQL scores range from 0-100 where higher scores indicate better health-related quality of life.
Time Frame: Baseline, 2 months, 3 months, 6 months, 9 months, 12 months post procedure
Population: The PEDsQL assessment is validated in patients under the age 18 years.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Occipital Nerve Block | Cervical Medial Branch Block
Number analyzed (Participants) | 3 | 3
units on a scale
  PedsQL Physical Functioning at Baseline | 53.1 [53.1 to 70.3] | 43.6 [40.6 to 68.8]
  PedsQL Emotional Functioning at Baseline | 75 [67.5 to 77.5] | 65 [60 to 82.5]
  PedsQL Social Functioning at Baseline | 100 [82.5 to 100] | 80 [67.5 to 90]
  PedsQL School Functioning at Baseline | 35 [30 to 50] | 55 [42.5 to 65]
  PedsQL Physical Functioning at 2 months: number analyzed (Participants) | 1 | 1
  PedsQL Physical Functioning at 2 months | 68.6 [68.6 to 68.6] | 34.4 [34.4 to 34.4]
  PedsQL Emotional Functioning at 2 months: number analyzed (Participants) | 1 | 1
  PedsQL Emotional Functioning at 2 months | 85 [85 to 85] | 90 [90 to 90]
  PedsQL Social Functioning at 2 months: number analyzed (Participants) | 1 | 1
  PedsQL Social Functioning at 2 months | 95 [95 to 95] | 70 [70 to 70]
  PedsQL School Functioning at 2 months: number analyzed (Participants) | 1 | 1
  PedsQL School Functioning at 2 months | 35 [lower limit 35] | 30 [30 to 30]
  PedsQL Physical Functioning at 3 months: number analyzed (Participants) | 3 | 1
  PedsQL Physical Functioning at 3 months | 62.5 [57.8 to 81.3] | 40.6 [40.6 to 40.6]
  PedsQL Emotional Functioning at 3 months: number analyzed (Participants) | 3 | 1
  PedsQL Emotional Functioning at 3 months | 85 [85 to 85] | 65 [65 to 65]
  PedsQL Social Functioning at 3 months: number analyzed (Participants) | 3 | 1
  PedsQL Social Functioning at 3 months | 90 [85 to 95] | 60 [60 to 60]
  PedsQL School Functioning at 3 months: number analyzed (Participants) | 3 | 1
  PedsQL School Functioning at 3 months | 50 [37.5 to 72.5] | 40 [40 to 40]
  PedsQL Physical Functioning at 6 months: number analyzed (Participants) | 3 | 0
  PedsQL Physical Functioning at 6 months | 65.6 [50 to 82.8] |
  PedsQL Emotional Functioning at 6 months: number analyzed (Participants) | 3 | 0
  PedsQL Emotional Functioning at 6 months | 75 [72.5 to 87.5] |
  PedsQL Social Functioning at 6 months: number analyzed (Participants) | 3 | 0
  PedsQL Social Functioning at 6 months | 100 [95 to 100] |
  PedsQL Sleep Functioning at 6 months: number analyzed (Participants) | 3 | 0
  PedsQL Sleep Functioning at 6 months | 50 [47.5 to 75] |
  PedsQL Physical Functioning at 9 months: number analyzed (Participants) | 3 | 1
  PedsQL Physical Functioning at 9 months | 65.6 [64.1 to 82.8] | 65.6 [65.6 to 65.6]
  PedsQL Emotional Functioning at 9 months: number analyzed (Participants) | 3 | 1
  PedsQL Emotional Functioning at 9 months | 100 [80 to 100] | 80 [80 to 80]
  PedsQL Social Functioning at 9 months: number analyzed (Participants) | 3 | 1
  PedsQL Social Functioning at 9 months | 100 [90 to 100] | 80 [80 to 80]
  PedsQL School Functioning at 9 months: number analyzed (Participants) | 3 | 1
  PedsQL School Functioning at 9 months | 50 [45 to 75] | 80 [80 to 80]
  PedsQL Physical Functioning at 12 months: number analyzed (Participants) | 1 | 1
  PedsQL Physical Functioning at 12 months | 100 [100 to 100] | 84.4 [84.4 to 84.4]
  PedsQL Emotional Functioning at 12 months: number analyzed (Participants) | 1 | 1
  PedsQL Emotional Functioning at 12 months | 100 [100 to 100] | 80 [80 to 80]
  PedsQL Social Functioning at 12 months: number analyzed (Participants) | 1 | 1
  PedsQL Social Functioning at 12 months | 100 [100 to 100] | 85 [85 to 85]
  PedsQL School Functioning at 12 months: number analyzed (Participants) | 1 | 1
  PedsQL School Functioning at 12 months | 100 [100 to 100] | 75 [75 to 75]

ADVERSE EVENTS:
Time Frame: Self-reported side effect data collected through surveys administered over a 12-month time period evaluated after study termination.
Description: Self-reported side effect data collected through surveys administered over a 12-month time period and Counts reflect the number of patients reporting side effect at least once. Data must be interpreted with caution due to longitudinal data collection design which may reflect results that are unrelated to the study.
Groups:
- Occipital Nerve Block_Initial Treatment: This arm/group represents the total number of patients who were randomized to the occipital nerve block treatment at the start of the study.
- Cervical Medial Branch Block_Initial Treatment: This arm/group represents the total number of patients who were randomized to the cervical medial branch block treatment at the start of the study.
- Crossover to CMBB From Initial ONB: This arm/group represents the total number of patients who were initially randomized to the occipital nerve block treatment at the start of the study but then crossed over to the cervical medial branch block treatment arm.
- Crossover to ONB From Initial CMBB: This arm/group represents the total number of patients who were initially randomized to the cervical medial branch block treatment at the start of the study but then crossed over to the occipital nerve block treatment arm.
Arm/Group | Occipital Nerve Block_Initial Treatment | Cervical Medial Branch Block_Initial Treatment | Crossover to CMBB From Initial ONB | Crossover to ONB From Initial CMBB
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 3/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Occipital Nerve Block_Initial Treatment (N=8) | Cervical Medial Branch Block_Initial Treatment (N=8) | Crossover to CMBB From Initial ONB (N=3) | Crossover to ONB From Initial CMBB (N=2)
Pain at the site of injection (Surgical and medical procedures) | 5 | 6 | 2 | 2
Bleeding from the site of injection (Surgical and medical procedures) | 1 | 0 | 0 | 0
Infection (warmth, redness, swelling) at the site of injection (Surgical and medical procedures) | 0 | 0 | 0 | 0
Neck stiffness (Surgical and medical procedures) | 7 | 8 | 3 | 2
Muscle soreness/pain (Surgical and medical procedures) | 7 | 8 | 3 | 2
Dizziness (Surgical and medical procedures) | 5 | 6 | 1 | 2
Upper limb numbness/weakness (Surgical and medical procedures) | 3 | 3 | 1 | 1
Fatigue (Surgical and medical procedures) | 7 | 7 | 2 | 2
Gait instability or balance problems (Surgical and medical procedures) | 2 | 5 | 1 | 2
Difficulty swallowing (Surgical and medical procedures) | 0 | 3 | 0 | 0
Other (Surgical and medical procedures) | 3 | 2 | 1 | 0

LIMITATIONS AND CAVEATS:
Even though post-traumatic headache management is multimodal, we have limited evidence of any current treatment options showing longer term benefits. The trial was preliminary halted due to difficulties with patient recruitment. As such, limited results have been presented which should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03007420/Prot_SAP_000.pdf